CLINICAL TRIAL: NCT04349267
Title: A Phase 1/2 Study of BMS-986315 as Monotherapy and in Combination With Nivolumab or Cetuximab in Participants With Advanced Solid Tumors
Brief Title: Study of BMS-986315 Alone and in Combination With Nivolumab or Cetuximab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA047-004
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: NSCLC (Non-small cell lung cancer); RCC (Renal cell carcinoma); SCCHN (Squamous cell carcinoma of the head and neck)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — Nivolumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986315 (Experimental)
  Interventions: Biological: BMS-986315
- BMS-986315 + nivolumab (Experimental)
  Interventions: Biological: BMS-986315; Biological: nivolumab
- BMS-986315 + cetuximab (Experimental)
  Interventions: Biological: BMS-986315; Biological: cetuximab

INTERVENTIONS:
Biological: BMS-986315 — Specified dose on specified days
Biological: nivolumab — Specified dose on specified days
  Arms: BMS-986315 + nivolumab
Biological: cetuximab — Specified dose on specified days
  Arms: BMS-986315 + cetuximab

SUMMARY:
The purpose of this study is to evaluate BMS-986315 alone and in combination with nivolumab or cetuximab in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic confirmation of advanced (metastatic, recurrent, and/or unresectable) squamous cell carcinoma of the head and neck (SCCHN), nonsmall cell lung cancer (NSCLC), or renal cell cancer (RCC) with measurable disease per RECIST 1.1
* Participants expected to have received standard of care therapies including an available PD-(L)1 inhibitor
* Eastern cooperative oncology group performance status of 0 or 1
* Women of childbearing potential must agree to follow methods of contraception

Exclusion Criteria:

* Participants with active, known or suspected autoimmune disease
* Participants with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
* Uncontrolled or significant cardiovascular disease
* History of or with active interstitial lung disease or pulmonary fibrosis
* Prior participation in anti-natural killer cell receptor (anti-NKG2A) clinical study
* History of allergy or hypersensitivity to study drug components

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (2):
  - Local Institution - 0028, Sioux Falls, South Dakota
  - Local Institution - 0001, Germantown, Tennessee
- Canada (5):
  - Local Institution - 0014, Edmonton, Alberta
  - Local Institution - 0011, Vancouver, British Columbia
  - Local Institution - 0004, Toronto, Ontario
  - Local Institution - 0005, Montreal, Quebec
  - Local Institution - 0013, Ottawa
- Local Institution, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Part 1C.
Groups:
- Part 1A BMS-986315-80 mg: Participants with select advanced tumors like Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC) and Non-small cell lung cancer (NSCLC) received 80 mg once in 4 weeks (Q4W) intravenously.
- Part 1A BMS-986315-200 mg: Participants with select advanced tumors like Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC) and Non-small cell lung cancer (NSCLC) received 200 mg once in 4 weeks (Q4W) intravenously.
- Part 1A BMS-986315-600 mg: Participants with select advanced tumors like Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC) and Non-small cell lung cancer (NSCLC) received 600 mg once in 4 weeks (Q4W) intravenously.
- Part 1A BMS-986315-1200 mg: Participants with select advanced tumors like Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC) and Non-small cell lung cancer (NSCLC) received 1200 mg once in 4 weeks (Q4W) intravenously.
- Part 1B BMS-986315-200 mg + Nivolumab 480 mg: Participants with select advanced tumors like Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC) and Non-small cell lung cancer (NSCLC) received 200 mg once in 4 weeks (Q4W) intravenously and Nivolumab 480 mg Q4W intravenously.
- Part 1B BMS-986315-600 mg + Nivolumab 480 mg: Participants with select advanced tumors like Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC) and Non-small cell lung cancer (NSCLC) received 600 mg once in 4 weeks (Q4W) intravenously and Nivolumab 480 mg Q4W intravenously.
- Part 1B BMS-986315-1200 mg + Nivolumab 480 mg: Participants with select advanced tumors like Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC) and Non-small cell lung cancer (NSCLC) received 1200 mg once in 4 weeks (Q4W) intravenously and Nivolumab 480 mg Q4W intravenously.
Period: Overall Study
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Started | 2 | 2 | 3 | 3 | 5 | 14 | 15
Completed | 0 | 0 | 1 | 0 | 1 | 5 | 3
Not Completed | 2 | 2 | 2 | 3 | 4 | 9 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other reason | 0 | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Disease Progression | 2 | 0 | 2 | 3 | 3 | 7 | 10
Not completed — Participant withdrew consent | 0 | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg | Total
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 14 | 15 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (18.38) | 68.5 (2.12) | 65.0 (9.00) | 63.0 (13.00) | 70.8 (6.91) | 67.4 (9.71) | 61.1 (8.93) | 64.9 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 1 | 6 | 6 | 16
  Male | 0 | 1 | 3 | 3 | 4 | 8 | 9 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2 | 3 | 4 | 11 | 10 | 32
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 1 | 3 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Black or African American | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 4
  White | 2 | 1 | 3 | 1 | 4 | 12 | 12 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Deaths
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition occurring in a clinical investigation participant after signing of informed consent, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory test result), symptom, or disease temporally associated with the study intervention. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose (Day 1) and 100 days after last dose of study therapy (up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 14 | 15
Participants
  Any adverse events | 2 | 2 | 3 | 3 | 5 | 14 | 15
  Serious Adverse Events | 0 | 2 | 0 | 0 | 3 | 8 | 10
  AEs leading to discontinuation | 0 | 1 | 0 | 0 | 0 | 2 | 2
  Deaths | 1 | 1 | 0 | 0 | 1 | 2 | 4

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A Dose Limiting Toxicity (DLT) is a treatment-related adverse event that is severe enough to prevent an increase in dose or continuation of therapy. DLTs include specific hepatic, hematologic, dermatologic, and other toxicities, such as Grade 4 liver enzyme elevations, Grade 4 cytopenias, persistent Grade 3 rashes, or serious organ toxicities unresponsive to treatment. Certain Grade 3 events (e.g., transient nausea, electrolyte imbalances) are excluded if they resolve quickly or with standard care.
Time Frame: From first dose (Day 1) untill Day 28
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 14 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants whose best overall response (BOR) is either CR or PR per response evaluation criteria in solid tumors (RECIST) v1.1 based on Clopper-Pearson method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of randomization to the date of first objectively documented progression or death, whichever occurs first (up to approximately 25 months)
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 14 | 15
percentage of participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 52.2] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8]

4. Secondary Outcome: Duration of Response (DoR)
Description: DOR for a participant with a best overall response (BOR) of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death, whichever occurs first. Median computed using Kaplan-Meier method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 3
Population: All treated participants. Only confirmed responders (CR or PR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
months |  |  |  |  |  | NA [NA to NA] — Median was not reached due to insufficient number of participants with events" and "95% CI not calculable for a single participant |

5. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: Progression Free Survival Rates at 6 months is defined as the percentage of participants who achieve PFS at 6 months. PFS for a participant is defined as the time from randomization date to the date of first objectively documented disease progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death due to any cause, whichever occurs first. Based on Kaplan-Meier Estimates.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: At 6 months
Population: All treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 14 | 15
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of BMS-986315
Description: Blood samples were collected to assess pharmacokinetic (PK) parameters.
Time Frame: Cycle 1 Day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 11 | 13
ug/mL | 28.8519 (40) | 51.9309 (13) | 168.2658 (3) | 283.6735 (66) | 63.1812 (15) | 160.8894 (35) | 309.0469 (24)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of BMS-986315
Description: Blood samples were collected to assess pharmacokinetic (PK) parameters.
Time Frame: Cycle 1 Day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 11 | 13
hours | 2.1916 (168) | 2.5151 (84) | 1.0747 (10) | 1.8572 (104) | 1.4213 (63) | 3.5165 (249) | 1.9030 (78)

8. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) of BMS-986315
Description: Blood samples were collected to assess pharmacokinetic (PK) parameters.
Time Frame: Cycle 1 Day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 11 | 13
h*ug/mL | 6885.1959 (33) | 12122.1650 (18) | 41381.3449 (12) | 62500.0455 (56) | 12885.5705 (20) | 36893.5416 (32) | 62110.3402 (33)

9. Secondary Outcome: Area Under the Concentration-time Curve in One Dosing Interval (AUC[Tau]) of BMS-986315
Description: Blood samples were collected to assess pharmacokinetic (PK) parameters.
Time Frame: Cycle 1 Day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 11 | 13
h*ug/mL | 6345.4606 (21) | 13113.1903 (6) | 41381.3449 (12) | 62500.0455 (56) | 12885.5705 (20) | 36893.5416 (32) | 70405.3800 (29)

10. Secondary Outcome: Concentration in a Dosing Interval (Ctau) of BMS-986315
Description: Blood samples were collected to assess pharmacokinetic (PK) parameters.
Time Frame: Cycle 1 Day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 5 | 11 | 13
ug/mL | 4.4119 (20) | 10.7013 (23) | 33.1011 (4) | 51.1321 (66) | 10.5418 (26) | 28.3387 (40) | 49.2124 (48)

11. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: An ADA positive participant was defined as participant with at least one ADA-positive sample relative to baseline (ADA negative at baseline or ADA titer to be at least 4-fold or greater (>=) than baseline positive titer) at any time after initiation of treatment.
Time Frame: Cycle 1 Day 1
Population: All treated participants with baseline and at least one post-baseline evaluable ADA assessment. Participants in Part 1A did not have at least one post-baseline evaluable assessment, hence no participants are included in analysis of Part1A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 12 | 12
Participants
  BMS986315 ADA |  |  |  |  | 0 | 0 | 0
  Nivolumab ADA |  |  |  |  | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from first dose Day 1 and up to approximately 49 months. Serious and Other Adverse events were collected from first dose (Day 1) and 100 days after last dose of study therapy (up to approximately 25 months).
Description: All-cause mortality, serious and other adverse events were collected for all the treated participants.
Arm/Group | Part 1A BMS-986315-80 mg | Part 1A BMS-986315-200 mg | Part 1A BMS-986315-600 mg | Part 1A BMS-986315-1200 mg | Part 1B BMS-986315-200 mg + Nivolumab 480 mg | Part 1B BMS-986315-600 mg + Nivolumab 480 mg | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/2 | 3/3 | 2/3 | 4/5 | 7/14 | 14/15
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/2 | 0/3 | 0/3 | 3/5 | 8/14 | 10/15
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 3/3 | 3/3 | 4/5 | 14/14 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A BMS-986315-80 mg (N=2) | Part 1A BMS-986315-200 mg (N=2) | Part 1A BMS-986315-600 mg (N=3) | Part 1A BMS-986315-1200 mg (N=3) | Part 1B BMS-986315-200 mg + Nivolumab 480 mg (N=5) | Part 1B BMS-986315-600 mg + Nivolumab 480 mg (N=14) | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 1 | 2
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
VIth nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A BMS-986315-80 mg (N=2) | Part 1A BMS-986315-200 mg (N=2) | Part 1A BMS-986315-600 mg (N=3) | Part 1A BMS-986315-1200 mg (N=3) | Part 1B BMS-986315-200 mg + Nivolumab 480 mg (N=5) | Part 1B BMS-986315-600 mg + Nivolumab 480 mg (N=14) | Part 1B BMS-986315-1200 mg + Nivolumab 480 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 5
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Saliva altered (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 2 | 9 | 5
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 2 | 0 | 3 | 4
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 3 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Bladder dilatation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 4 | 4
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT04349267/Prot_SAP_000.pdf